CLINICAL TRIAL: NCT05004714
Title: Implementation of a Multilevel Program to Reduce Asthma Symptoms in Urban Preschoolers
Brief Title: Y of Central Maryland Head Start Asthma Implementation
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00244099; R01HL146785-01A1 (NIH)
Record Dates: First submitted 2021-08-11; First posted 2021-08-13 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Asthma in Children; Implementation; Preschool Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Head Start Staff: Head Start staff including teachers, family advocates, directors, and others
- Head Start Children with Asthma: Children enrolled in Head Start program with physician diagnosed asthma

SUMMARY:
Despite a strong evidence-base for the efficacy of multilevel programs in reducing asthma symptoms among low-income preschool minority children, gaps remain in our understanding of how to best translate and scale up these efficacious interventions into sustainable programs that reduce known asthma health disparities. Head Start (HS) serves over one million low income children in the US each year by focusing on early learning, physical health, and family engagement. HS is committed to implementing evidence based programs to promote overall child well-being, and is focused on addressing asthma symptoms due to the deleterious impact on school absences and child development. We have demonstrated the effectiveness of a multi-level staff and family education program (ABC Asthma) that significantly reduced asthma symptoms and courses of oral corticosteroids. However, these interventions are not successfully integrated within community organizations for long-term sustainability. It is unknown how to best scale up and implement these evidence based asthma interventions into low resource community organizations that serve children at risk. Implementation strategies are frequently developed atheoretically and may not be tailored to the setting. The overall purpose of this project is to inform best practices of implementation of an asthma education program by 1) systematically evaluating the use of intervention mapping to develop a tailored implementation strategy in partnership with Head Start stakeholders, 2) examining both staff and organizational level determinants associated with implementation of ABC Asthma, and 3) evaluating the success of tailored implementation strategies on implementation outcomes and school absences and other health outcomes. The YMCA of Central Maryland have enthusiastically agreed to implement the Maryland ABC HS Asthma within 40 sites in four communities: Baltimore City, Baltimore County, Anne Arundel County, and Prince George's County.

ELIGIBILITY:
Aim 1

Inclusion Criteria:

* Aged 18 or older
* Head Start Staff member or caregiver of child currently enrolled in Head Start with asthma
* Cognitive ability to provide consent
* Willing to be audio recorded

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Head Start Staff member or caregiver of child currently enrolled in Head Start with asthma
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
School Absences due to asthma symptoms | 5 years
  Child Level Outcome

SECONDARY OUTCOMES:
Implementation evaluation | 5 years
  Adoption and penetration

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Eakin, PhD, Principal Investigator — JHU
Locations (2):
- United States (2):
  - Easter Seals Head Start Prince George's County, District Heights, Maryland
  - Y of Central Maryland Head Start, Nottingham, Maryland

IPD SHARING:
Plan to Share IPD: No